CLINICAL TRIAL: NCT02945800
Title: Phase II Study of Nab-Paclitaxel in Combination With Gemcitabine for Treatment of Recurrent/Refractory Sarcoma in Teenagers and Young Adults
Brief Title: Nab-Paclitaxel and Gemcitabine for Recurrent/Refractory Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Pediatric Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-18613
Record Dates: First submitted 2016-10-25; First posted 2016-10-26 (Estimated); Results first posted 2025-12-01 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Osteosarcoma; Ewing Sarcoma; Rhabdomyosarcoma; Soft Tissue Sarcoma
Keywords: relapsed; refractory; soft tissue; bones and joints; non-rhabdomyosarcoma soft tissue sarcoma; pediatric
MeSH Terms: conditions — Osteosarcoma; Sarcoma, Ewing; Rhabdomyosarcoma; Sarcoma; Recurrence | interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Combination Therapy (Experimental): Participants will receive nab-Paclitaxel and Gemcitabine on days 1, 8, and 15 of each 28 day cycle, for up to 12 cycles.
  Interventions: Drug: nab-Paclitaxel; Drug: Gemcitabine

INTERVENTIONS:
Drug: nab-Paclitaxel — nab-Paclitaxel: 125 mg/m^2 intravenously (IV)
  Other Names: Abraxane
Drug: Gemcitabine — Gemcitabine: 1000 mg/m^2 intravenously (IV)
  Other Names: Gemzar

SUMMARY:
The purpose of this study is to see if nab-paclitaxel combined with gemcitabine prevents the formation or growth of tumors in participants with relapsed or refractory osteosarcoma, Ewing sarcoma, rhabdomyosarcoma and other soft tissue sarcoma and to measure the length of time during and after treatment that their disease does not get worse. Researchers also want to find out if nab-paclitaxel combined with gemcitabine is safe and tolerable.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be age ≥ 3 and ≤ 30 years, and have had a histologic diagnosis of osteosarcoma, Ewing sarcoma, or rhabdomyosarcoma or non-rhabdomyosarcoma soft tissue sarcoma either at diagnosis or relapse. Must have experienced relapse after front-line therapy, or have had documented disease progression during front-line therapy.
* Must have measurable disease that can be assessed using Response Evaluation in Solid Tumors (RECIST) 1.1, defined as the presence of at least one lesion on MRI or CT scan that can be accurately measured with the longest diameter of 10 mm in at least one dimension. For this phase II trial, patients with disease limited to bone or marrow metastases are NOT eligible, as disease at these sites cannot be assessed by RECIST 1.1 criteria.
* Must have relapsed or refractory cancers for which there is no known curative option.
* Prior Therapy: There is no limit to the number of prior therapies provided all eligibility criteria are met. However, participants must have recovered from the acute toxic effects of all prior treatment. (A) Must not have received prior therapy with either gemcitabine or nab-paclitaxel. (B) Myelosuppressive chemotherapy: Must not have received myelosuppressive chemotherapy within 3 weeks of protocol therapy on this study. (C) Hematopoietic growth factors: 7 days must have elapsed from the start of protocol therapy since the completion of therapy with filgrastim, and 14 days must have elapsed from the start of protocol therapy after receiving pegfilgrastim. (D) Biologic (anti-neoplastic agent): 7 day must have elapsed from the start of protocol therapy since the completion of therapy with a biologic agent. (E) Monoclonal antibodies: 3 half-lives must have elapsed from the start of protocol therapy since prior therapy that included a monoclonal antibody. (F) Radiotherapy: 2 weeks must have elapsed from the start of protocol therapy since local palliative radiotherapy (small port); 3 months must have elapsed if 50% radiation of pelvis; 6 weeks must have elapsed if other substantial bone marrow irradiation was given. (G) Stem Cell Transplant or Rescue: No evidence of active graft vs. host disease and 2 months must have elapsed from the start of protocol therapy since transplant.
* Karnofsky performance score must be ≥ 60
* Must have organ and marrow function
* Neuropathy: Must have ≤ grade 1 neuropathy at enrollment
* Central nervous system (CNS) Metastases: Potential participants with known CNS metastases are excluded unless treated surgically or with radiotherapy and stable with no recurrent lesions for at least 3 months from the start of protocol therapy.
* Contraception: Women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation. Men treated or enrolled on this protocol must also agree to use adequate contraception 4 months after completion of gemcitabine and nab-paclitaxel administration.
* Consent: Participants must have the ability to understand and the willingness to sign a written informed consent or assent document.

Exclusion Criteria:

* Potential participants who are receiving any other investigational agents
* Must not be receiving any additional medicines being given for the specific purpose of treating cancer
* A history of allergic reactions attributed to docetaxel or paclitaxel
* Concomitant Medications: The metabolism of paclitaxel is catalyzed by CYP2C8 and CYP3A4. The following medicines should be avoided on this study because of their ability to inhibit or induce with CYP2C8 or CYP3A4: A) Inhibitors: ketoconazole and other imidazole antifungals, erythromycin, fluoxetine, gemfibrozil, cimetidine, ritonavir, saquinavir, indinavir, and nelfinavir. B) Inducers: Rifampicin, carbamazepine, phenytoin, efavirenz, and nevirapine. C) Potential participants receiving any of the above medications are ineligible.
* Potential participants are ineligible if they have uncontrolled intercurrent illness including, but not limited to: ongoing or active infection; symptomatic congestive heart failure; unstable angina pectoris; cardiac arrhythmia; psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or breastfeeding
* HIV Infection: HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with the study medications.
* Anyone who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study.

Ages: 3 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 59 (Actual)
Dates: Start 2016-10-25 (Actual); Primary Completion 2024-11-19 (Actual); Study Completion 2025-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Javier E. Oesterheld, M.D., Principal Investigator — Carolinas Medical Center, Levine Cancer Institute
Locations (14):
- United States (14):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Children's Hospital Los Angeles, Los Angeles, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - A.I. duPont Hospital for Children, Delaware - Nemours, Wilmington, Delaware
  - Shand's Hospital for Children at the University of Florida, Gainesville, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - Holtz Children's Hospital at the University of Miami, Miami, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Coordinating Center, Tampa, Florida
  - University of Kentucky, Lexington, Kentucky
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Carolinas Medical Center, Levine Cancer Institute, Charlotte, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - Vanderbilt - Ingram Cancer Center, Nashville, Tennessee

REFERENCES:
- [Derived] Hattinger CM, Patrizio MP, Magagnoli F, Luppi S, Serra M. An update on emerging drugs in osteosarcoma: towards tailored therapies? Expert Opin Emerg Drugs. 2019 Sep;24(3):153-171. doi: 10.1080/14728214.2019.1654455. Epub 2019 Aug 14. PMID 31401903
- See also: Moffitt Cancer Center Clinical Trials website — https://moffitt.org/clinical-trials-research/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Combination Therapy
Started | 59
Completed | 59
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Combination Therapy
Number analyzed (Participants) | 59
Age, Continuous [Mean (Full Range); unit: years] | 18.7 [8 to 30]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 44
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 13
  White | 34
  More than one race | 0
  Unknown or Not Reported | 9
Region of Enrollment [Number; unit: participants]
  United States | 59

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Treatment response will be assessed with the most relevant imaging studies (e.g., CT or MRI) after every two cycles. Standard Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 will be used to assess responses. Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm (<1 cm). Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: 13 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Combination Therapy
Number analyzed (Participants) | 59
percentage of participants | 15.3 [7.2 to 27.0]

2. Primary Outcome: Progression Free Survival (PFS)
Description: Progression-free survival (PFS) is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first. Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm (0.5 cm).
Time Frame: 13 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Combination Therapy
Number analyzed (Participants) | 59
Months | 1.91 [1.64 to 4.21]

3. Secondary Outcome: Occurrence of Study Treatment Related Adverse Events
Description: Adverse Events (AEs) and Serious Adverse Events (SAEs) according to Common Terminology Criteria for Adverse Events (CTCAE) V4.0, deemed to be caused by study treatment.
Time Frame: 13 months
Population: A total of 54 out of 59 patients experienced at least one event related to the study treatment.
Measure: Number; unit: participants
Arm/Group | Combination Therapy
Number analyzed (Participants) | 59
participants | 54

ADVERSE EVENTS:
Time Frame: 13 Months
Arm/Group | Combination Therapy
All-Cause Mortality (participants affected / at risk) | 24/59
Serious Adverse Events (participants affected / at risk) | 35/59
Other Adverse Events (participants affected / at risk) | 58/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Therapy (N=59)
Anemia (Blood and lymphatic system disorders) | 7 (7)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (6)
Sinus tachycardia (Cardiac disorders) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 3 (3)
Fatigue (General disorders) | 1 (2)
Fever (General disorders) | 15 (18)
Localized edema (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 3 (3)
Esophageal infection (Infections and infestations) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 2 (2)
Lung infection (Infections and infestations) | 2 (2)
Skin infection (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 1 (1)
Neutrophil count decreased (Investigations) | 3 (4)
Platelet count decreased (Investigations) | 5 (6)
Dehydration (Metabolism and nutrition disorders) | 4 (4)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hypotension (Vascular disorders) | 5 (5)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2)
Edema limbs (General disorders) | 3 (3)
Pain (General disorders) | 8 (9)
Sepsis (Infections and infestations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2)
Headache (Nervous system disorders) | 1 (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Vascular disorders - Other, specify (Vascular disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Therapy (N=59)
Neutrophil count decreased (Investigations) | 36 (75)
Platelet count decreased (Investigations) | 34 (82)
White blood cell decreased (Investigations) | 33 (60)
Lymphocyte count decreased (Investigations) | 28 (48)
Alanine aminotransferase increased (Investigations) | 10 (14)
Aspartate aminotransferase increased (Investigations) | 5 (5)
Alkaline phosphatase increased (Investigations) | 2 (2)
Blood bilirubin increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Investigations - Other, specify (Investigations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 36 (68)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (6)
Fever (General disorders) | 14 (16)
Fatigue (General disorders) | 6 (7)
Pain (General disorders) | 5 (6)
Non-cardiac chest pain (General disorders) | 4 (5)
Edema limbs (General disorders) | 3 (5)
Localized edema (General disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 6 (8)
Nausea (Gastrointestinal disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Mucositis oral (Gastrointestinal disorders) | 2 (3)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 9 (10)
Peripheral motor neuropathy (Nervous system disorders) | 5 (6)
Headache (Nervous system disorders) | 2 (2)
Syncope (Nervous system disorders) | 2 (2)
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 (10)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 2 (3)
Lung infection (Infections and infestations) | 2 (2)
Skin infection (Infections and infestations) | 2 (2)
Tooth Infection (Infections and infestations) | 2 (2)
Esophageal infection (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 6 (7)
Dehydration (Metabolism and nutrition disorders) | 4 (4)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 4 (6)
Pericardial effusion (Cardiac disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Hypertension (Vascular disorders) | 3 (3)
Hypotension (Vascular disorders) | 3 (3)
Thromboembolic event (Vascular disorders) | 1 (1)
Vascular disorders - Other, specify (Vascular disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-03): https://cdn.clinicaltrials.gov/large-docs/00/NCT02945800/Prot_SAP_000.pdf